CLINICAL TRIAL: NCT02565602
Title: A Comparative Study of Calcium Metabolism in Caucasian and Asian Postmenopausal Women of Chinese Descent and the Use of Strontium as a Qualitative Marker of Calcium Metabolism in Humans
Brief Title: Comparison of Calcium Metabolism in Caucasian and Asian Postmenopausal Women of Chinese Descent and the Use of Strontium as a Qualitative Marker of Calcium Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Thomas Walczyk, Associate Professor, National University of Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012/01000
Record Dates: First submitted 2015-09-21; First posted 2015-10-01 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Calcium Metabolism
Keywords: Calcium metabolism; Osteoporosis; Postmenopausal women
MeSH Terms: conditions — Osteoporosis | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ca-41 & Sr-84 (isotope tracers) & vit D (Other): Dosages: 3.7 kBq (100 nCi) Ca-41, 5 mg of Sr-84 and 400IU of vitamin D (daily)
  Interventions: Other: Ca-41(isotope tracer); Other: Sr-84 (isotope tracer); Dietary Supplement: Vitamin D

INTERVENTIONS:
Other: Ca-41(isotope tracer) — Ca-41 is given orally in the form of (Ca-41)Cl3 in citrate-buffered solution. Tracer will be used to determine parameters of calcium metabolism based on tracer excretion data.
Other: Sr-84 (isotope tracer) — Sr-84 is given orally in the form of (Sr-84)Cl2 in aqueous solution.Tracer will be used to determine parameters of strontium metabolism based on tracer excretion data.
Dietary Supplement: Vitamin D — One tablet daily (400IU per tablet)
  Other Names: Cholecalciferol

SUMMARY:
This study aims to: 1) quantitatively assess parameters of bone calcium balance in healthy postmenopausal Asian women of Chinese descent; 2) assess possible ethnic differences in calcium metabolism by direct comparison of acquired data in Chinese postmenopausal women with those acquired earlier in Caucasian postmenopausal women using the same methodology; 3) assess differences in calcium and strontium metabolism in parallel to evaluate if strontium stable isotopes can be used for tracing bone calcium metabolism qualitatively

DETAILED DESCRIPTION:
The study will follow closely the protocol that was used previously by the PI at ETH Zurich to study calcium metabolism in healthy postmenopausal women. Calcium metabolism will be studied after a single oral administration of a calcium tracer (Ca-41) and by following the excretion of the tracer in urine over 6 months. Obtained data will be used to assess parameters of calcium metabolism (flux rates and sizes of body calcium compartments) by kinetic modelling. A strontium tracer (Sr-84) will be administered in parallel and its urinary excretion pattern compared to Ca-41 excretion to determine if strontium tracers can be used to assess calcium metabolism qualitatively. Subjects will be supplemented with Vit D throughout the study. Vit D supplementation will commence 1 month before isotope administration.

ELIGIBILITY:
Inclusion Criteria:

1. Last menstrual bleeding was at least 5 years ago.
2. Between the ages of 50 and 75 years old.
3. Both parents and 4 grandparents are/were of Chinese descent. It is not a necessity for the participant, participant's parents and grandparent's to be born and raised in Singapore to participate in this study.
4. BMI above 16 and below 30

Exclusion Criteria:

1. Diagnosed with osteoporosis
2. Presence of significant liver disease, malignancy (excluding myeloma in the study group), malabsorption syndrome, hypoparathyroidism, hyperparathyroidism, sarcoidosis or hyperthyroidism (from toxic multinodular goitre or Graves disease), Paget's disease osteosarcoma, acromegaly, Cushing's syndrome, hypopituitarism, diabetes mellitus or severe chronic obstructive pulmonary disease.
3. Current smoking and an alcohol intake exceeding one standard drink per day
4. Undergoing treatment with any of the following drugs (within the last 12 months) i) adrenocorticoid steroids (3 months or longer at anytime or >10 days of treatment within the previous 12 months) ii) anticonvulsant therapy iii) pharmacological doses of thyroid hormone (causing decline of TSH below normal) iv) bisphosphonates v) calcitonin vi) synthetic parathyroid hormone vii) selective estrogen receptor modulators viii) strontium ranelate ix) estrogen therapy x ) chemotherapeutic agents xi) sodium fluoride (any history of treatment with fluoride) xii) medications known to affect calcium metabolism (diuretics, antacids, calcium channel blockers etc.).
5. Presence of any other chronic illnesses.
6. Any other significant medical, psychiatric and/or social issue as determined by the investigator that would compromise subject's safety and/or compliance with trial procedure.
7. Any other clinically significant screening laboratory abnormality (as determined by the investigators).

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Time changes in urinary tracer excretion (Ca-41 and Sr-84) | 6 months post dose
  Urine samples collected from participants are analysed for calcium and strontium content as well as Ca-41 and Sr-84 excretion.

SECONDARY OUTCOMES:
Flux rates and relative compartment sizes (mineralized bone, exchangeable bone calcium, plasma calcium) of the study population | 6 months post dose
  Flux rates (mg/day) and calcium distribution between compartments (% body calcium) will be obtained by compartmental modelling of urinary tracer data. Obtained data will be compared to a mirroring study conducted earlier in Caucasian postmenopausal women.
Comparison between flux rates and relative compartment sizes for calcium and strontium in each individual subject | 6 months post dose
  Flux rates (mg/day), and calcium and strontium distribution between compartments (% body calcium and strontium ) will be obtained by compartmental modelling of urinary tracer data

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Walczyk, Principal Investigator — National University of Singapore; Lawrence Lee, Principal Investigator — National University Health System
Locations (1):
- Investigational Medicine Unit, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Cabrera WE, Schrooten I, De Broe ME, D'Haese PC. Strontium and bone. J Bone Miner Res. 1999 May;14(5):661-8. doi: 10.1359/jbmr.1999.14.5.661. No abstract available. PMID 10320513
- [Background] Denk E, Hillegonds D, Vogel J, Synal A, Geppert C, Wendt K, Fattinger K, Hennessy C, Berglund M, Hurrell RF, Walczyk T. Labeling the human skeleton with 41Ca to assess changes in bone calcium metabolism. Anal Bioanal Chem. 2006 Nov;386(6):1587-602. doi: 10.1007/s00216-006-0795-5. Epub 2006 Oct 11. PMID 17033771
- [Background] Denk E, Hillegonds D, Hurrell RF, Vogel J, Fattinger K, Hauselmann HJ, Kraenzlin M, Walczyk T. Evaluation of 41calcium as a new approach to assess changes in bone metabolism: effect of a bisphosphonate intervention in postmenopausal women with low bone mass. J Bone Miner Res. 2007 Oct;22(10):1518-25. doi: 10.1359/jbmr.070617. PMID 17576167
- [Background] Lee WH, Wastney ME, Jackson GS, Martin BR, Weaver CM. Interpretation of 41Ca data using compartmental modeling in post-menopausal women. Anal Bioanal Chem. 2011 Feb;399(4):1613-22. doi: 10.1007/s00216-010-4454-5. Epub 2010 Dec 9. PMID 21152905
- [Background] Lin Y, Hillegonds DJ, Gertz ER, Van Loan MD, Vogel JS. Protocol for assessing bone health in humans by tracing long-lived 41Ca isotope in urine, serum, and saliva samples. Anal Biochem. 2004 Sep 1;332(1):193-5. doi: 10.1016/j.ab.2004.05.019. No abstract available. PMID 15301966
- [Background] Suzuki T. Risk factors for osteoporosis in Asia. J Bone Miner Metab. 2001;19(3):133-41. doi: 10.1007/s007740170032. No abstract available. PMID 11368297
- [Background] Villegas R, Gao YT, Dai Q, Yang G, Cai H, Li H, Zheng W, Shu XO. Dietary calcium and magnesium intakes and the risk of type 2 diabetes: the Shanghai Women's Health Study. Am J Clin Nutr. 2009 Apr;89(4):1059-67. doi: 10.3945/ajcn.2008.27182. Epub 2009 Feb 18. PMID 19225116
- [Background] Wastney ME, Martin BR, Peacock M, Smith D, Jiang XY, Jackman LA, Weaver CM. Changes in calcium kinetics in adolescent girls induced by high calcium intake. J Clin Endocrinol Metab. 2000 Dec;85(12):4470-5. doi: 10.1210/jcem.85.12.7004. PMID 11134095
- [Background] Wu L, Martin BR, Braun MM, Wastney ME, McCabe GP, McCabe LD, DiMeglio LA, Peacock M, Weaver CM. Calcium requirements and metabolism in Chinese-American boys and girls. J Bone Miner Res. 2010 Aug;25(8):1842-9. doi: 10.1002/jbmr.76. PMID 20205166
- [Background] International Commission on Radiological Protection (1991) Biological aspects of radiological protection. Annals of the ICRP. 21, 11-25.
- [Background] Dose coefficients for intakes of radionuclides by workers. A report of a Task Group of Committee 2 of the International Commission on Radiological Protection. Ann ICRP. 1994;24(4):1-83. No abstract available. PMID 7668473
- [Background] Schulze-König, T., Maden, C., Denk, E., Freeman, S. P. H. T., Stocker, M., Suter, M., Synal, A., Walczyk, T. (2010) Comparison of 41Ca analysis on 0.5 MV and 5 MV-AMS systems. Nuclear Instruments and Methods in Physics Research B. 268, 752-755.